CLINICAL TRIAL: NCT02710136
Title: A Pilot Study to Assess Safety and Feasibility of Cockroach Nasal Allergen Challenge in Cockroach Sensitive Children and Adults With Asthma (ICAC-27)
Brief Title: Cockroach Nasal Allergen Challenge Pilot
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Inner-City Asthma Consortium (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAIT ICAC-27; CoNAC (Other: ICAC)
Record Dates: First submitted 2016-03-07; First posted 2016-03-16 (Estimated); Results first posted 2018-08-28 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-08

CONDITIONS: Asthma; Cockroach Hypersensitivity
Keywords: Asthma; Glycerinated German cockroach allergenic extract; Cockroach Nasal Allergen Challenge
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Glycerinated CR Allergenic Extract (Experimental): Complete Arm Title: Glycerinated German Cockroach Allergenic Extract.
  Cockroach sensitive subjects are exposed to cockroach nasal allergen (NAC) intranasally at at increasing doses per protocol. The NAC aim is pursuit of optimal dose range as determined by tolerability and eliciting a threshold of nasal symptoms.
  Interventions: Biological: Glycerinated German Cockroach Allergenic Extract

INTERVENTIONS:
Biological: Glycerinated German Cockroach Allergenic Extract — Participants will receive escalating doses intranasally. Briefly: per protocol- Phase 1a NAC: N=10 cockroach sensitive adults with asthma will undergo nasal allergen challenge with dose escalation (up to 8 doses per protocol). Phase 1b: Phase 1a subjects will have repeat NAC with dose escalation (up to 8 doses).
  Phase 2: N=25 cockroach sensitive children with asthma (ages 8 - 14 years) will undergo NAC with doses determined by Phase 1a data (e.g., symptoms and safety data).
  Other Names: Blattella germanica allergenic extract; Cockroach antigen (CR antigen)

SUMMARY:
This research is being done to look at the body's response to cockroach extract, an allergen, when sprayed into the nose. The spraying of the cockroach extract into the participant's nose is called Nasal Allergen Challenge (NAC). The purpose of this study is to evaluate the safety and tolerability of a intranasal cockroach extract given to participants with asthma.

DETAILED DESCRIPTION:
This is a multi-center, open label pilot study to assess the safety and determine the feasibility of cockroach nasal allergen challenge in children with asthma. This pilot study will occur in two phases:

* Phase 1 will enroll 10 cockroach sensitive adults with asthma who will undergo a nasal allergen challenge with increasing doses of cockroach allergen. Phase 1 will consist of two parts, Phase 1a and Phase 1b. In Phase 1a, participants will undergo a nasal allergen challenge. In Phase 1b, participants will undergo a repeat nasal allergen challenge to assess reproducibility of the NAC with cockroach allergen in a population with asthma. The data from Phase 1a will be used to identify a range of doses that is safe and elicits a threshold of nasal symptoms (TNSS ≥8).
* Phase 2 will enroll 25 cockroach sensitive children with asthma ages 8-14 years who will undergo a nasal allergen challenge using the dose range identified in Phase 1a.

Study mandated procedures include: blood draws (venipuncture); pulmonary function testing (PFTs); nasal allergen challenge (NAC); allergen skin testing; and peak expiratory flow.

ELIGIBILITY:
Accrual Objective: N=10 adults, 25 children)

STUDY INCLUSION CRITERIA:

* Subjects fulfilling all of the following criteria are eligible for enrollment as study participants for Phase 1a and Phase 2:

  1. Subject and/or parent guardian must be able to understand and provide informed consent.
  2. Male or female adults, 18 through 55 years of age at recruitment (Phase 1) or male or female children, 8-14 years of age at recruitment (Phase 2).
  3. Have a history of asthma for a minimum of 1 year before study entry:

     1. A diagnosis of asthma for this study is defined as a reported clinical diagnosis of asthma made by a physician over a year ago.
     2. The subject must have persistent asthma defined by the current need for at least 100 microgram (mcg) fluticasone per day or the equivalent of another inhaled corticosteroid.
     3. The subject's asthma must be well controlled as defined by:

        * A Forced Expiratory Volume in 1 Second (FEV1) ≥ 80% predicted.
        * An Asthma Control Test (ACT) score ≥ 20.
  4. Are sensitive to German Cockroach as documented by a positive (≥ 3 mm greater than negative control) skin prick test result and a positive German Cockroach specific immunoglobulin E (IgE) (≥0.35 kUA/L).
  5. Have no known contraindications to the allergenic extracts or diluents.
* Subjects who meet the following criteria are eligible for enrollment as study participants in Phase 1b after completion of Phase 1a:

  1. Their asthma must be well controlled as defined by:

     1. A FEV1 ≥ 80% predicted.
     2. An Asthma Control Test (ACT) score ≥ 20.
  2. The subject tolerated the Nasal Allergen Challenge (NAC) during Phase 1a with no adverse events grade 2 or higher as determined by "Guidance for Industry: Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials (published September 2007) for local reactions to study procedures."
* Subjects not eligible for enrollment as study participants in Phase 1b after completion of Phase 1a if any of the following criteria are met:

  1. Are pregnant or lactating.
  2. Have an asthma severity classification of severe persistent, using the NAEPP classification, as evidenced by at least one of the following:

     1. Require a dose of greater than 500 mcg of fluticasone per day or the equivalent of another inhaled corticosteroid.
     2. Have received more than 2 courses of oral or parenteral corticosteroids within the last 12 months or one course within the last 3 months.
     3. Have been treated with depot corticosteroids within the last 12 months.
     4. Have been hospitalized for asthma within the 12 months prior to their participation in Phase1b.
     5. Have had an emergency room visit for asthma within the 3 months prior to their participation in Phase 1b.
     6. Have had a life-threatening asthma exacerbation that required intubation, mechanical ventilation, or that resulted in a hypoxic seizure within 2 years prior to their participation in Phase 1b.
  3. Have received allergen immunotherapy (SLIT or SCIT) in the last 12 months prior to their participation in Phase 1b.
  4. Have previously been treated with anti-IgE therapy in the 12 months prior to their participation in Phase 1b.
  5. Are currently receiving oral or nasal antihistamines, nasal corticosteroids, nasal decongestants, nasal anticholinergics or cromolyn, which cannot be suspended for the required washout periods prior to the nasal allergen challenge in Phase 1b.
  6. Have received an investigational drug in the 30 days prior to their participation in Phase 1b.
  7. Have past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the subject's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study.
  8. Meet any of the Participant Stopping Rules and Withdrawal Criteria during Phase 1a

     * The participant elected to withdraw consent from all future study activities, including followup.
     * The Investigator no longer believes participation is in the best interest of the participant.
     * Serious Adverse Event (SAE) related to investigational product.
     * Anaphylactic reaction grade 2 or 3.
     * Inability to tolerate the NAC prior to reaching a TNSS ≥8 due to excessive discomfort or symptoms.
     * Epistaxis occurring during the Challenge Visit.
     * The need to start immunotherapy or any chronic immunosuppressive medications in the period between Phase 1a and Phase 1b.
     * Require a dose of greater than 500 mcg of fluticasone per day or the equivalent of another inhaled corticosteroid to maintain asthma control in the period between Phase 1a and Phase 1b.
     * Inability to restrict use of antihistamines, nasal steroids, nasal decongestants, nasal anticholinergics or cromolyn prior to the NAC.
     * Development of any serious medical illness whose natural history, sequela, or treatment would be worsened or impaired by continuation in the protocol.
     * Subject is "lost to follow-up"
  9. The subject's initial TNSS at the Repeat Challenge Visit must be within 1 point of the initial TNSS at the Challenge Visit in Phase 1a. If the participant's initial TNSS is outside the 1 point range, then the participant may be reevaluated for the Repeat Challenge Visit up to 3 additional times.

STUDY EXCLUSION CRITERIA:

Subjects fulfilling any of the following criteria are not eligible for enrollment in any portion of the study and may not be reassessed. Participants are ineligible if they:

1. Plan to move from the area during the study period.
2. Have a history of idiopathic anaphylaxis or anaphylaxis grade 2 or higher as defined by the grading scale of Brown et al. for anaphylaxis and systemic reactions to study procedures.
3. Have unstable angina, significant arrhythmia, uncontrolled hypertension, history of autoimmune disease, or other chronic or immunological diseases that in the opinion of the investigator might interfere with the evaluation of the investigational agent or pose additional risk to the participant.
4. Are using tricyclic antidepressants or beta-adrenergic blocker drugs (both oral and topical).

EXCLUSION CRITERIA SPECIFIC TO STUDY PHASE 1A AND -2:

* Subjects who meet any of these criteria are not eligible for enrollment as study participants in Phase1a and Phase 2:

  1. Are pregnant or lactating. Post-menarcheal females must be abstinent or use a medically acceptable birth control method throughout the study (e.g. oral, subcutaneous, mechanical, or surgical contraception).
  2. Cannot perform spirometry at Screening.
  3. Have an asthma severity classification at Recruitment of severe persistent, using the The National Asthma Education and Prevention Program (NAEPP) classification, as evidenced by at least one of the following:

     1. Require a dose of greater than 500mcg of fluticasone per day or the equivalent of another inhaled corticosteroid.
     2. Have received more than 2 courses of oral or parenteral corticosteroids within the last 12 months or one course within the last 3 months.
     3. Have been treated with depot corticosteroids within the last 12 months.
     4. Have been hospitalized for asthma within the 12 months prior to recruitment.
     5. Have had an emergency room visit for asthma within the 3 months prior to recruitment.
     6. Have had a life-threatening asthma exacerbation that required intubation, mechanical ventilation, or that resulted in a hypoxic seizure within 2 years prior to recruitment.
  4. Have nasal polyps or other major structural abnormalities in their nasal cavities as assessed by anterior rhinoscopy.
  5. Have active rhinitis symptoms prior to the nasal allergen challenge, defined as a Baseline Total Nasal Symptom Score(TNSS) >3,with no individual symptom score >1.
  6. Do not have access to a phone (needed for scheduling appointments).
  7. Have received allergen immunotherapy (Sublingual [SLIT] or Subcutaneous [SCIT]) in the last 12 months prior to recruitment or who plan to initiate or resume allergen immunotherapy during the study.
  8. Have previously been treated with anti-IgE therapy in the 12 months prior to recruitment.
  9. Are currently receiving oral or nasal antihistamines, nasal corticosteroids, nasal decongestants,nasal anticholinergics or cromolyn, which cannot be suspended for the required washout periods prior to skin prick testing and the nasal allergen challenge.
  10. Have received an investigational drug in the 30 days prior to recruitment or who plan to use an investigational drug during the study.
  11. Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study.

Ages: 8 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Actual)
Dates: Start 2016-02; Primary Completion 2017-04-11 (Actual); Study Completion 2017-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Wood, MD, Study Chair — Johns Hopkins University
Locations (4):
- United States (4):
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - UT Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
The plan is to share data upon completion of the study in ImmPort, a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts.
Time Frame: The aim is to share data available to the public within 24 months upon completion of the study.
Access Criteria: ImmPort public data access.
URL: http://www.immport.org/immport-open/public/home/home

REFERENCES:
- [Derived] Rudman Spergel AK, Sever ML, Johnson J, Gill MA, Schulten V, Frazier A, Kercsmar CM, Lovinsky-Desir S, Searing DA, Sette A, Shao B, Teach SJ, Gern JE, Busse WW, Togias A, Wood RA, Liu AH; National Institute of Allergy and Infectious Diseases Inner City Asthma Consortium. Development of nasal allergen challenge with cockroach in children with asthma. Pediatr Allergy Immunol. 2021 Jul;32(5):971-979. doi: 10.1111/pai.13480. Epub 2021 Mar 20. PMID 33606312
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 182 participants recruited, 80 participants consented to be screened for study eligibility. Among the five participating clinical research sites, all located in the United States, 35 participants enrolled to participate in the study. Enrollment was active from February 2016 to March 2017.
Groups:
- Cockroach Sensitive Adults With Asthma: In Phase 1a, adult participants ages 18-55 underwent a nasal allergen challenge (NAC) with increasing doses of German cockroach allergen. At each allergen dose, the Total Nasal Symptom Score (TNSS; 0-12) was determined. This score is the sum of subscale scores measuring sneezing (0-3), runny nose (0-3), stuffy nose (0-3), and itchy nose (0-3) symptoms. Results were used to identify a range of doses that are safe and elicit nasal symptoms of TNSS ≥8 or a sneezing score=3. Participants who completed the NAC in Phase 1a were invited to assess additional screening criteria and return for a second nasal allergen challenge in Phase 1b to evaluate the reproducibility of the NAC in determining nasal symptoms in response to German cockroach allergen.
- Cockroach Sensitive Children With Asthma: In Phase 2, pediatric participants ages 8-14 underwent a nasal allergen challenge with increasing doses of German cockroach allergen. At each allergen dose, the Total Nasal Symptom Score (TNSS; 0-12) was determined. This score is the sum of subscale scores measuring sneezing (0-3), runny nose (0-3), stuffy nose (0-3), and itchy nose (0-3) symptoms. Results were used to identify a range of doses that are safe and elicit nasal symptoms of TNSS ≥6 or a sneezing score=3.
Period: Study Enrollment
Arm/Group | Cockroach Sensitive Adults With Asthma | Cockroach Sensitive Children With Asthma
Started | 10 | 25
Completed | 10 | 25
Not Completed | 0 | 0
Period: Phase 1a[Refer to Arm/Group Description]
Arm/Group | Cockroach Sensitive Adults With Asthma | Cockroach Sensitive Children With Asthma
Started | 10 | 0
Completed | 9 | 0
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Phase 1b[Refer to Arm/Group Description]
Arm/Group | Cockroach Sensitive Adults With Asthma | Cockroach Sensitive Children With Asthma
Started | 4 | 0
Completed | 4 | 0
Not Completed | 0 | 0
Period: Phase 2 [Refer to Arm/Group Description]
Arm/Group | Cockroach Sensitive Adults With Asthma | Cockroach Sensitive Children With Asthma
Started | 0 | 25
Completed | 0 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Phase 1a and Phase 2 participants who started a Nasal Allergen Challenge
Groups:
- Total: Total of all reporting groups
Arm/Group | Cockroach Sensitive Adults With Asthma | Cockroach Sensitive Children With Asthma | Total
Number analyzed (Participants) | 10 | 25 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 25 | 25
  Between 18 and 65 years | 10 | 0 | 10
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.0 (7.5) | 11.2 (1.9) | 15.5 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 3 | 16 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 6 | 6
  Not Hispanic or Latino | 10 | 19 | 29
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 18 | 28
  White | 0 | 6 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 25 | 35
German cockroach allergen Bla g 1, Bla g 2, or Bla g 5 ng/g levels in home dust above LLD (yes/no) [Count of Participants; unit: Participants] — Blatella germanica 1 (Bla g 1), Blatella germanica 2 (Bla g 2), and Blatella germanica 5 (Bla g 5) are cockroach proteins that cause allergy to cockroach in humans. Levels above the lower limit of detection (LLD) indicate the presence of cockroaches in the home. LLD for Bla g 1, Bla g 2, and Bla g 5 were 120, 196, and 140 ng/g, respectively.
  Participants | 1 | 9 | 10
German cockroach allergen skin test wheal size (mm) [Geometric Mean (Standard Deviation); unit: mm] — Extent of allergy to German cockroach can be assessed using a skin prick test. In this test, a small amount of allergen is introduced to the skin via a needle, and then the diameter of the resulting swelling, called a wheal, is measured. Larger wheal sizes indicate greater allergy to German cockroach.
  mm | 6.2 (1.6) | 5.6 (1.5) | 5.8 (1.5)
German cockroach allergen IgE (kU/L) [Geometric Mean (Standard Deviation); unit: kU/L] — Extent of allergy to German cockroach can be assessed using levels of German cockroach specific Immunoglobulin E (IgE). IgE are antibodies produced by the immune system, so that higher levels of IgE present indicate greater allergy to German cockroach. IgE levels are measured in the serum (blood test).
  kU/L | 3.61 (4.60) | 3.48 (4.61) | 3.52 (4.50)
Total Nasal Symptom Score (TNSS) [Mean (Standard Deviation); unit: Scores on a Scale] — Total Nasal Symptom Score (TNSS) (0-12) is a participant rated score computed as the sum of four subscale scores (0-3) measuring sneezing, runny nose, stuffy nose, and itchy nose symptoms. Participants indicate a score on each subscale of 0, 1, 2, or 3, indicating none, mild, moderate, or severe symptoms, respectively. Baseline TNSS scores were obtained after the nasal rinse administered prior to the Nasal Allergen Challenge. Higher scores indicate more severe nasal symptoms.
  Scores on a Scale | 0.50 (0.71) | 1.04 (1.06) | 0.89 (0.99)
Peak Nasal Inspiratory Flow (PNIF) L/min [Mean (Standard Deviation); unit: L/min] — PNIF is defined as the speed of inspiration of air in Liters per minute when breathing into the lungs. Baseline PNIF scores were obtained after the nasal rinse administered prior to the Nasal Allergen Challenge. Lower scores indicate less ability to breathe air into the lungs due to more severe nasal symptoms.
  L/min | 150.5 (36.1) | 108.8 (37.8) | 120.7 (41.4)
Peak Expiratory Flow (PEF) L/min [Mean (Standard Deviation); unit: L/min] — PEF is defined as the speed of expiration of air in Liters per minute when breathing out of the lungs. Baseline PEF scores were obtained after the nasal rinse administered prior to the Nasal Allergen Challenge. Lower scores indicate less ability to expel air out of the lungs due to more severe nasal symptoms.
  L/min | 362.5 (103.3) | 303.0 (88.9) | 320.0 (95.6)
Visual Analog Score (VAS) [Mean (Standard Deviation); unit: Centimeters] — Participants self-reported their score, reflecting the severity of their nasal symptoms-sneezing, runny nose, stuffy nose, itchy nose- on a Visual Analogue Scale (0 to 10 centimeters). The left-hand side of the scale (0) represents "No Symptoms," and the right hand side of the scale (10) represents "As Bad as I Can Imagine." Baseline VAS scores were obtained after the nasal rinse administered prior to the Nasal Allergen Challenge.
  Centimeters | 0.12 (0.26) | 1.07 (1.88) | 0.80 (1.64)
Log base 10 Tryptase in Nasal Secretions [Mean (Standard Deviation); unit: mcg/L] — Tryptase is a protein in the human body whose levels are hypothesized to be related to extent of allergic response. Baseline tryptase scores were obtained after the nasal rinse administered prior to the Nasal Allergen Challenge. Higher scores indicate more allergic response.
  mcg/L | 0.49 (0.69) | 0.84 (0.73) | 0.71 (0.72)
Log base 10 Albumin in Nasal Secretions [Mean (Standard Deviation); unit: mcg/L] — Albumin is a protein in the human body whose levels are hypothesized to be related to extent of allergic response. Baseline albumin scores were obtained after the nasal rinse administered prior to the Nasal Allergen Challenge. Higher scores indicate more allergic response.
  mcg/L | 5.39 (0.69) | 5.80 (0.44) | 5.67 (0.55)

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Proportion of Participants Meeting Either a Total Nasal Symptom Score (TNSS) Threshold or Sneezing Score Threshold During the Cockroach Allergen (CA) Nasal Allergen Challenge (NAC)
Description: Result is the proportion of participants (Pss) responding at each of 9 CA doses during the NAC.To illustrate the variability of the outcome at each dose,the protocol specifies computation of 95% CIs for the proportion responding at each dose.A proportion is to record for each Ps a 0 for non-responder and 1 for responder &compute the mean of the 0 &1 values.Summary statistic for this method: a mean.
  After each dose,TNSS &TNSS Sneezing scores were recorded.TNSS (0-12) is a self-rated score computed as the sum of 4 subscale scores (0-3) measuring sneezing, runny nose, stuffy nose, & itchy nose symptoms (sxs).Pss provide a score on each subscale of 0, 1, 2, or 3(none, mild, moderate, or severe sxs, respectively).Pss cont'd receiving doses until either a TNSS (≥8 in adults,≥6 in children) or sneezing score threshold [TLV] of 3 was met.Assumption: Pss met TLV criteria for doses not recv'd beyond dose at which TLV criteria were initially met.
Time Frame: NAC Baseline through last dose of German cockroach allergen administered during the NAC
Population: Phase 1a and Phase 2 Participants who started a NAC
Measure: Mean (95% Confidence Interval); unit: Cumulative proportion of participants
Arm/Group | Cockroach Sensitive Adults With Asthma | Cockroach Sensitive Children With Asthma
Number analyzed (Participants) | 10 | 25
Cumulative proportion of participants
  Dose 1 - 0 mcg/mL | 0.00 [0.00 to 0.31] | 0.12 [0.03 to 0.31]
  Dose 2 - 0.00381 mcg/mL | 0.00 [0.00 to 0.31] | 0.16 [0.05 to 0.36]
  Dose 3 - 0.01204 mcg/mL | 0.10 [0.00 to 0.45] | 0.16 [0.05 to 0.36]
  Dose 4 - 0.0380 mcg/mL | 0.22 [0.03 to 0.60] | 0.32 [0.15 to 0.54]
  Dose 5 - 0.120 mcg/mL | 0.44 [0.14 to 0.79] | 0.48 [0.28 to 0.69]
  Dose 6 - 0.379 mcg/mL | 0.56 [0.21 to 0.86] | 0.64 [0.43 to 0.82]
  Dose 7 - 1.20 mcg/mL | 0.56 [0.21 to 0.86] | 0.72 [0.51 to 0.88]
  Dose 8 - 3.78 mcg/mL | 0.56 [0.21 to 0.86] | 0.76 [0.55 to 0.91]
  Dose 9 - 11.9 mcg/mL | 0.67 [0.30 to 0.93] | 0.80 [0.59 to 0.93]

2. Secondary Outcome: Number of Sneezes at Each of Nine Doses of German Cockroach Allergen
Description: Nine increasing doses of German cockroach allergen (0, 0.00381, 0.01204, 0.0380, 0.120, 0.379, 1.20, 3.78, and 11.9 mcg/mL) were administered during the Nasal Allergen Challenge (NAC). After administration of each dose, the number of times the participant sneezed was recorded. Participants continued receiving doses of German cockroach allergen until threshold criteria described in the primary endpoint were met. Number of sneezes was carried forward for doses not received beyond the dose at which the threshold criteria were initially met. Number of sneezes is summarized at each dose.
Time Frame: NAC Baseline through last dose of German cockroach allergen administered during the NAC
Population: Phase 1a and Phase 2 Participants who started a NAC
Measure: Mean (Standard Deviation); unit: Count of sneezes
Arm/Group | Cockroach Sensitive Adults With Asthma | Cockroach Sensitive Children With Asthma
Number analyzed (Participants) | 10 | 25
Count of sneezes
  Dose 1 - 0 mcg/mL | 0.00 (0.00) | 0.32 (0.99)
  Dose 2 - 0.00381 mcg/mL | 0.00 (0.00) | 0.76 (1.64)
  Dose 3 - 0.01204 mcg/mL | 0.50 (0.97) | 0.64 (1.41)
  Dose 4 - 0.0380 mcg/mL | 1.40 (2.55) | 1.56 (2.48)
  Dose 5 - 0.120 mcg/mL | 3.10 (3.63) | 2.80 (3.62)
  Dose 6 - 0.379 mcg/mL | 3.80 (4.42) | 4.04 (4.61)
  Dose 7 - 1.20 mcg/mL | 4.00 (4.27) | 4.20 (4.49)
  Dose 8 - 3.78 mcg/mL | 4.10 (4.23) | 4.48 (4.48)
  Dose 9 - 11.9 mcg/mL | 4.40 (4.25) | 4.68 (4.36)

3. Secondary Outcome: Highest Total Nasal Symptom Score (TNSS)
Description: TNSS (0-12) is a participant rated score computed as the sum of four subscale scores (0-3) measuring sneezing, runny nose, stuffy nose, and itchy nose symptoms. Participants provide a score on each subscale of 0, 1, 2, or 3, indicating none, mild, moderate, or severe symptoms, respectively. The highest TNSS observed after administration of any of the German cockroach allergen doses received during the Nasal Allergen Challenge (NAC) is summarized.
Time Frame: NAC Baseline through last dose of German cockroach allergen administered during the NAC
Population: Phase 1a and Phase 2 Participants who started a NAC
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Cockroach Sensitive Adults With Asthma | Cockroach Sensitive Children With Asthma
Number analyzed (Participants) | 10 | 25
Scores on a Scale | 5.20 (3.05) | 5.16 (2.12)

4. Secondary Outcome: Change in Total Nasal Symptom Score (TNSS)
Description: TNSS (0-12) is a participant rated score computed as the sum of four subscale scores (0-3) measuring sneezing, runny nose, stuffy nose, and itchy nose symptoms. Participants indicate a score on each subscale of 0, 1, 2, or 3, indicating none, mild, moderate, or severe symptoms, respectively. Change is computed by subtracting the TNSS score obtained after the nasal rinse administered prior to the Nasal Allergen Challenge from the TNSS score obtained at the last tolerated dose of German cockroach allergen received during the Nasal Allergen Challenge (NAC). A positive change score indicates that nasal symptoms increased over the course of the NAC.
Time Frame: NAC Baseline through last dose of German cockroach allergen administered during the NAC
Population: Phase 1a and Phase 2 Participants who started a NAC
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Cockroach Sensitive Adults With Asthma | Cockroach Sensitive Children With Asthma
Number analyzed (Participants) | 10 | 25
Scores on a Scale | 4.40 (3.17) | 3.96 (2.35)

5. Secondary Outcome: Change in Peak Nasal Inspiratory Flow (PNIF) L/Min
Description: PNIF is defined as the speed of inspiration of air in Liters per minute when breathing into the lungs. Change is computed by subtracting the PNIF score obtained after the nasal rinse administered prior to the Nasal Allergen Challenge (NAC) from the PNIF score obtained at the last tolerated dose of German cockroach allergen received during the NAC. A negative change score indicates that speed of inspiration decreased over the course of the NAC.
Time Frame: NAC Baseline through last dose of German cockroach allergen administered during the NAC
Population: Phase 1a and Phase 2 Participants who started a NAC
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Cockroach Sensitive Adults With Asthma | Cockroach Sensitive Children With Asthma
Number analyzed (Participants) | 10 | 25
L/min | -33.5 (44.5) | -18.8 (34.0)

6. Secondary Outcome: Change in Peak Expiratory Flow (PEF) L/Min
Description: PEF is defined as the speed of expiration of air in Liters per minute when breathing out of the lungs. Change is computed by subtracting the PEF score obtained after the nasal rinse administered prior to the Nasal Allergen Challenge (NAC) from the PEF score obtained at the last tolerated dose of German cockroach allergen received during the NAC. A positive change score indicates that speed of expiration increased over the course of the Challenge, while a negative change score indicates speed of expiration decreased over the course of the NAC.
Time Frame: NAC Baseline through last dose of German cockroach allergen administered during the NAC
Population: Phase 1a and Phase 2 Participants who started a NAC
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Cockroach Sensitive Adults With Asthma | Cockroach Sensitive Children With Asthma
Number analyzed (Participants) | 10 | 25
L/min | 25.0 (57.0) | -5.2 (27.4)

7. Secondary Outcome: Change in Visual Analogue Score
Description: Participants self-reported their score, reflecting the severity of their nasal symptoms-sneezing, runny nose, stuffy nose, itchy nose- on a Visual Analogue Scale (0 to 10 centimeters). The left-hand side of the scale (0) represents "No Symptoms," and the right hand side of the scale (10) represents "As Bad as I Can Imagine."
  Change is computed by subtracting the VAS score obtained after the nasal rinse administered prior to the Nasal Allergen Challenge (NAC) from the VAS score obtained at the last tolerated dose of German cockroach allergen received during the NAC. A positive change score indicates that nasal symptoms increased over the course of the NAC.
Time Frame: NAC Baseline through last dose of German cockroach allergen administered during the NAC
Population: Phase 1a and Phase 2 Participants who started a NAC
Measure: Mean (Standard Deviation); unit: Centimeters
Arm/Group | Cockroach Sensitive Adults With Asthma | Cockroach Sensitive Children With Asthma
Number analyzed (Participants) | 10 | 25
Centimeters | 1.82 (1.66) | 1.44 (1.92)

8. Secondary Outcome: Change in Log Base 10 Tryptase in Nasal Secretions
Description: Tryptase is a protein in the human body. Levels are hypothesized to be related to the extent of allergic response. Change is computed by subtracting the tryptase level prior to the Nasal Allergen Challenge (NAC) from the tryptase level after the last dose received during the NAC. A log base 10 transformation is applied to both baseline and post-baseline measures. A positive change score indicates that tryptase levels increased over the course of the NAC.
Time Frame: NAC Baseline through last dose of German cockroach allergen administered during the NAC
Population: Phase 1a and Phase 2 Participants who started a NAC and had an evaluable baseline and post-baseline tryptase measurement.
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | Cockroach Sensitive Adults With Asthma | Cockroach Sensitive Children With Asthma
Number analyzed (Participants) | 10 | 17
mcg/L | 0.55 (0.52) | 0.25 (0.63)

9. Secondary Outcome: Change in Log Base 10 Albumin in Nasal Secretions
Description: Albumin is a protein in the human body. Levels are hypothesized to be related to the extent of allergic response. Change is computed by subtracting the albumin level prior to the Nasal Allergen Challenge (NAC) from the albumin level after the last dose received during the NAC. A log base 10 transformation is applied to both baseline and post-baseline measures. A positive change score indicates that albumin levels increased over the course of the NAC.
Time Frame: NAC Baseline through last dose of German cockroach allergen administered during the NAC
Population: Phase 1a and Phase 2 Participants who started a NAC and had an evaluable baseline and post-baseline albumin measurement.
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | Cockroach Sensitive Adults With Asthma | Cockroach Sensitive Children With Asthma
Number analyzed (Participants) | 10 | 17
mcg/L | 0.32 (0.61) | 0.19 (0.35)

ADVERSE EVENTS:
Time Frame: Time of consent until participant completed study participation or until 10 days have participant prematurely withdraws (without withdrawing consent) or was withdrawn from the study
Groups:
- Phase 1a Cockroach Sensitive Adults With Asthma: Adverse events captured during Screening and Phase 1a are included. In Phase 1a, adult participants ages 18-55 underwent a nasal allergen challenge (NAC) with increasing doses of German cockroach allergen. At each allergen dose, the Total Nasal Symptom Score (TNSS; 0-12) was determined. This score is the sum of subscale scores measuring sneezing (0-3), runny nose (0-3), stuffy nose (0-3), and itchy nose (0-3) symptoms. Results were used to identify a range of doses that are safe and elicit nasal symptoms of TNSS ≥8 or a sneezing score=3. Participants who completed the NAC in Phase 1a were invited to return for a second nasal allergen challenge in Phase 1b to assess the reproducibility of the NAC in determining nasal symptoms in response to German cockroach allergen.
- Phase 1b Cockroach Sensitive Adults With Asthma: Adverse events captured during Phase 1b are included. In Phase 1a, adult participants ages 18-55 underwent a nasal allergen challenge (NAC) with increasing doses of German cockroach allergen. At each allergen dose, the Total Nasal Symptom Score (TNSS; 0-12) was determined. This score is the sum of subscale scores measuring sneezing (0-3), runny nose (0-3), stuffy nose (0-3), and itchy nose (0-3) symptoms. Results were used to identify a range of doses that are safe and elicit nasal symptoms of TNSS ≥8 or a sneezing score=3. Participants who completed the NAC in Phase 1a were invited to assess additional screening criteria and return for a second nasal allergen challenge in Phase 1b to evaluate the reproducibility of the NAC in determining nasal symptoms in response to German cockroach allergen.
- Cockroach Sensitive Children With Asthma: Adverse events captured during Phase 2 are included. In Phase 2, pediatric participants ages 8-14 underwent a nasal allergen challenge with increasing doses of German cockroach allergen. At each allergen dose, the Total Nasal Symptom Score (TNSS; 0-12) was determined. This score is the sum of subscale scores measuring sneezing (0-3), runny nose (0-3), stuffy nose (0-3), and itchy nose (0-3) symptoms. Results were used to identify a range of doses that are safe and elicit nasal symptoms of TNSS ≥6 or a sneezing score=3.
Arm/Group | Phase 1a Cockroach Sensitive Adults With Asthma | Phase 1b Cockroach Sensitive Adults With Asthma | Cockroach Sensitive Children With Asthma
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/4 | 0/25
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/4 | 1/25
Other Adverse Events (participants affected / at risk) | 4/10 | 2/4 | 7/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1a Cockroach Sensitive Adults With Asthma (N=10) | Phase 1b Cockroach Sensitive Adults With Asthma (N=4) | Cockroach Sensitive Children With Asthma (N=25)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1a Cockroach Sensitive Adults With Asthma (N=10) | Phase 1b Cockroach Sensitive Adults With Asthma (N=4) | Cockroach Sensitive Children With Asthma (N=25)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0)
Vessel puncture site pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Xerosis (General disorders) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Peak expiratory flow rate decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (3) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-09-09): https://cdn.clinicaltrials.gov/large-docs/36/NCT02710136/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-06): https://cdn.clinicaltrials.gov/large-docs/36/NCT02710136/SAP_001.pdf